CLINICAL TRIAL: NCT02661295
Title: The Effect of Ferric Citrate on Inflammation and Lipid Levels in Patients on Hemodialysis
Brief Title: A Study of Ferric Citrate to Improve Inflammation and Lipid Levels
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 38 enrolled, 19 completed the study when loss of funding occurred
Sponsor: Winthrop University Hospital (Other)
Collaborators: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WUH 756275-1
Record Dates: First submitted 2016-01-11; First posted 2016-01-22 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: End Stage Renal Disease; Hyperphosphatemia; Chronic Inflammation
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — ferric citrate

STUDY DESIGN:
Intervention Model Description: This study will be designed as a single arm, prospective, experimental trial of 45 hemodialysis patients. Patients on hemodialysis at least 6 months and receiving a phosphate binder with serum phosphorus levels between 2.5 and 8.0 mg/dL, normal serum calcium levels, and on maintenance iron therapy are potentially eligible. Participants will receive ferric citrate after at least a 2 week washout period from previous phosphate binders if phosphorus is ≥ 5.5 mg/dl, calcium is within the normal range and ferritin ≥ 200 and < 600 ng/ml. Ferric citrate will be titrated to maintain serum phosphorus and calcium within acceptable levels. Inflammatory markers and lipid levels will be tested at 0, 3, and 6 months.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferric Citrate (Other): Ferric citrate at a starting dose of 2 tablets with each meal will be given to all participants.
  Interventions: Drug: Ferric Citrate

INTERVENTIONS:
Drug: Ferric Citrate — Study participants will receive ferric citrate at a starting dose of 2 tablets with each meal if serum phosphorus levels are ≥ 6.0 mg/dL calcium levels are in the normal range, Tsat ≥ 20 and < 50% and ferritin ≥ 200 and < 500 ng/ml after a 2 week wash out period.
  Other Names: Auryxia

SUMMARY:
The risk of cardiovascular mortality in patients with end stage renal disease on hemodialysis is 10-100 times higher than the normal population. This is due in part to high levels of inflammation and vascular calcification found in these patients. Phosphate binders, particularly non-calcium based phosphate binders, may decrease cardiovascular risk by decreasing inflammation and vascular calcification. Ferric citrate a non-calcium based phosphate binder with approximately 210 mg of ferric iron has recently been approved for patients on hemodialysis. The effect of this phosphate binder on inflammation and lipid levels is unknown but investigators hypothesize that ferric citrate has the potential to improve inflammation and lipid levels in patients on hemodialysis by decreasing intravenous iron requirements and by improving lipid metabolism.

DETAILED DESCRIPTION:
In patients with end stage renal disease (ESRD) receiving dialysis, the risk of cardiovascular death has been estimated to be 10-100 times higher than the general population without renal disease. This is due in part to high levels of inflammation and vascular calcification (large deposits of calcium in arteries) found in these patients. Chronic inflammation is particularly common in patients with ESRD. Parenteral iron therapy, which is common in patients on dialysis, may contribute to this inflammation and also a higher cardiovascular risk. Phosphate binders, particularly non-calcium based phosphate binders, may decrease cardiovascular risk by decreasing inflammation and vascular calcification. In a study of 10,044 hemodialysis patients, treatment with a phosphate binder was associated with improved survival. Ferric citrate a non-calcium based phosphate binder with approximately 210 mg of ferric iron has recently been approved for patients on hemodialysis. It has been shown to improve serum phosphorus levels and decrease intravenous iron requirements for patients on hemodialysis. The effect of this phosphate binder on inflammation and lipid levels is unknown but investigators hypothesize that ferric citrate has the potential to improve inflammation and lipid levels in patients on hemodialysis by decreasing intravenous iron requirements and by improving lipid metabolism.

Ferric citrate has the potential to decrease cardiovascular risk through multiple mechanisms:

1. acting as a non-calcium based binder to decrease serum phosphorus levels and vascular calcification,
2. decreasing intravenous iron requirements which in turn may decrease inflammation,
3. binding endotoxin (a harmful substance produced by microorganisms) in the gut and
4. improving lipid metabolism.

The purpose of this study is to examine the effect of ferric citrate on inflammatory markers and lipid levels.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis treatment for ≥ 6 months
* Phosphate binder treatment for ≥ to 1 month
* Maintenance iron therapy with no more than 125mg IV iron weekly≥ to 1 month
* Serum phosphorus levels between 2.5 and 8 at screening
* Serum phosphorus ≥ to 6.0 mg/dL after a 2 week washout period.
* Serum ferritin ≥ 200 and < 600ng/ml after a 2 week washout period
* Serum calcium levels within normal range
* Predicted survival greater than 6 months

Exclusion Criteria:

* Intact PTH< 70 pg/ml or > 1,000 pg/ml
* Oral iron use
* Vitamin C supplement use
* Parathyroidectomy
* Active malignancy
* Hemodialysis via an intravenous catheter or arteriovenous (AV) graft
* Received > 250mg of IV iron over the two weeks prior to screening
* Whole blood transfusion within 3 months prior to screening
* Active bleeding other than from the dialysis access
* Hospitalization within one month prior to screening
* current infection
* Ongoing or uncontrolled inflammatory disorder
* Liver cirrhosis
* Likelihood of imminent renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09-29 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace Grant, MD, Principal Investigator — NYU Winthrop
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferric Citrate
Started | 38
Completed | 19
Not Completed | 19
Not completed — Death | 1
Not completed — Transferred Out | 1
Not completed — Kidney Transplant | 1
Not completed — Withdrawn due to side effects | 8
Not completed — Withdrawn due to access type | 1
Not completed — Withdrawn due to allergies | 1
Not completed — Withdrawn due to non-compliance | 1
Not completed — Withdrawal by Subject | 3
Not completed — Failed screening | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Cholesterol
Description: Percent change in total cholesterol (mg/dl) from Baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | 1.58 (33.77)

2. Primary Outcome: Percent Change in LDL-Cholesterol
Description: Percent change in low-density lipoprotein (LDL) cholesterol (mg/dl) from baseline to Month 6
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | -0.05 (32.47)

3. Primary Outcome: Percent Change in HDL Cholesterol
Description: Percent change in high-density lipoprotein (HDL) cholesterol (mg/dl) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | 1.32 (6.16)

4. Primary Outcome: Percent Change in Triglycerides
Description: Percent change in triglycerides (mg/dl) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | -5.11 (67.69)

5. Primary Outcome: Percent Change in TNF-alpha
Description: Percent change in tumor necrosis factor (TNF)-alpha (pg/ml) from Baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | -0.1 (1.77)

6. Primary Outcome: Percent Change in IL-6
Description: Percent change in interleukin 6 (IL-6) (pg/ml) from baseline to Month 6
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | -1.78 (19.5)

7. Primary Outcome: Percent Change in IL-8
Description: Percent change in interleukin 8 (IL-8) (pg/ml) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | 101.96 (422.8)

8. Primary Outcome: Percent Change in Ferritin
Description: Percent change in ferritin (ng/ml) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | 51.11 (296.4)

9. Primary Outcome: Percent Change in C-reactive Protein
Description: Percent change in C-reactive Protein (mg/L) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | 8.89 (35.49)

10. Primary Outcome: Percent Change in Homocysteine
Description: Percent change in homocysteine (micromol/L) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
percent change | 1.35 (7.31)

11. Primary Outcome: Change in Intravenous Iron Use
Description: Change in intravenous iron use (mg) from Baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
mg | -588.8 (807.8)

12. Secondary Outcome: Percent Change in Calcium
Description: Percent change in calcium (mg/dL) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | 0.08 (0.53)

13. Secondary Outcome: Percent Change in Phosphorus
Description: Percent change in phosphorus (md/dl) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | -1.58 (1.87)

14. Secondary Outcome: Percent Change in Parathyroid Hormone (PTH)
Description: Percent change in PTH (pg/ml) from baseline to Month 6.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 19
Percent change | 36.47 (280.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ferric Citrate
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Citrate (N=38)
Renal transplant (Renal and urinary disorders) | 1
Coronary artery bypass graft (Cardiac disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Encephalomalacia (Nervous system disorders) | 1
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Fluid overload (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lethargy (Nervous system disorders) | 1
Chest pain (General disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Catheter infection (Product Issues) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT02661295/Prot_SAP_000.pdf